CLINICAL TRIAL: NCT04854291
Title: A Randomized, Double Blind, Placebo Controlled Multicenter Trial of Fecal Microbiome Transplantation Safety and Efficacy for Parkinson's Disease Patients with Abnormal Gut Microbiota Composition
Brief Title: A Trial of Fecal Microbiome Transplantation in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Tampere University Hospital (Other); University of Helsinki (Other); Central Hospital of Paijat-Hame (Unknown); University of Aarhus (Other)
Responsible Party: Principal Investigator, Filip Scheperjans, Adjunct Professor of Neurology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD-FMT
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; FMT; microbiota; gut-brain axis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donor FMT (Experimental): FMT from a healthy donor
  Interventions: Other: Administration of donor FMT
- Placebo (Placebo Comparator): NaCl + glycerol mixture (carrier solution of FMT arm)
  Interventions: Other: Administration of placebo

INTERVENTIONS:
Other: Administration of donor FMT — Intracaecal infusion of FMT
  Arms: Donor FMT
Other: Administration of placebo — Intracaecal infusion of carrier solution
  Arms: Placebo

SUMMARY:
48 PD patients (age 35-75y; H&Y 1-3) testing positive in a stool PD-dysbiosis test will be randomized in a 2:1 ratio to receive either donor FMT or their own stool through intracaecal infusion. The main outcome measure will be the sum of MDS-UPDRS I-III at 6 months to cover motor and non-motor symptom changes. A wide array of secondary clinical outcome measures will be assessed longitudinally and a large array of measurements, biospecimens (stool, urine, blood, colonic biopsies), and imaging data will be collected for further analysis at baseline, 1, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD (Clinically Probable PD)
* H&Y OFF 1-3 at Baseline Visit

Exclusion Criteria:

1. Chronic gastrointestinal disease (IBS allowed, celiac disease allowed if on gluten free diet, gastritis allowed)
2. Any previous major gastrointestinal surgery that may alter gastrointestinal physiology
3. Any abdominal surgery in the last 3 months
4. Major genital and/or rectum prolapse
5. Active autoimmune disease
6. Active cancer within 5 years (allowed: basalioma and successfully removed carcinoma in situ)
7. Immune deficiency
8. HIV infection
9. Antibiotic use in last 3 months before baseline visit
10. Dementia as indicated by Moca <21p
11. Psychosis
12. Active significant impulse control disorder (by interview and medical records)
13. Major depression as indicated by BDI-II >28
14. Pregnancy
15. Alcohol or drug abuse
16. Negative dysbiosis test result
17. Iodine allergy
18. Deep brain stimulation or Duodopa/Lecigon treatment
19. Inability to interrupt regular use of NSAIDs for at least one month before permeability assessments

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Change of the sum of MDS-UPDRS I-III from baseline | at 6 months post intervention
  Sum of Movement Disorder Society Unified Parkinson's Disease Rating Scale sum of parts I, II, and III (in OFF state); Min 0 - Max 236 points (higher points indicating worse symptoms) will be determined at baseline and at 6 months after intervention. The difference between these values will be the primary outcome measure; Min 0 - Max 236 points (higher points indicating stronger improvement)

SECONDARY OUTCOMES:
Change of MDS-UPDRS III from baseline | at 6 and 12 months post intervention
  Movement Disorder Society Unified Parkinson's Disease Rating Scale part III (in OFF state); Min 0 - Max 132 points (higher points indicating worse symptoms) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 132 points (higher points indicating stronger improvement)
Change of MDS-UPDRS IV from baseline | at 6 and 12 months post intervention
  Movement Disorder Society Unified Parkinson's Disease Rating Scale part IV; Min 0 - Max 132 points (higher points indicating worse symptoms) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 24 points (higher points indicating stronger improvement)
Change of Timed UP GO test from baseline | at 6 and 12 months post intervention
  measured in seconds, higher value indicating worse clinical symptoms expressed as difference between 6 and 12 month post intervention and baseline, higher value indicating stronger improvement
Change of MDS-UPDRS I from baseline | at 6 and 12 months post intervention
  Movement Disorder Society Unified Parkinson's Disease Rating Scale part I; Min 0 - Max 52 points (higher points indicating worse symptoms) will be determined at baseline and at 6 months after intervention. The difference between these values will be calculated; Min 0 - Max 52 points (higher points indicating stronger improvement)
Change of NMSS from baseline | at 6 and 12 months post intervention
  Non-motor symptom scale (0-360 points, higher points indicating worse symptoms) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 360 points (higher points indicating stronger improvement)
Change in gut permeability, motility and volume from baseline | at 6 months
  Gut permability is studied using the Iohexole test.Motility and volume is studied using radio-opaque markers and volume measurments from abdominal CT scans
Change of fecal and blood markers from baseline | whole study period
  Shotgun metagenomics based taxonomic microbiota survey, metabolomics, inflammatory markers, DNA methylation
Change of BDI-II from baseline | at 6 and 12 months post intervention
  Beck Depression Inventory II (0-63 points, higher points indicating worse symptoms) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 63 points (larger decrease indicating stronger improvement)
Change of BAI from baseline | at 6 and 12 months post intervention
  Beck Anxiety inventory will be determined at baseline and at 6 and 12 months after intervention.
  The difference between these values will be calculated; Min 0 - Max 63 points (larger decrease indicating stronger improvement)
Change of RBDSQ from baseline | at 6 and 12 months after intervention
  REM sleep behavior disorder screening questionnaire will be determined at baseline and at 6 and 12 months after intervention.
Change of MoCa from baseline | at 6 and 12 months post intervention
  MONTREAL COGNITIVE ASSESSMENT (0-30 points, higher points indicating less symptoms) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 30 points (higher increase indicating stronger improvement)
Change of IBS-SSS from baseline | at 6 and 12 months after intervention
  The irritable bowel severity scoring system will be determined at baseline and follow-up
Change of PDQ39 index from baseline | at 6 and 12 months post intervention
  Parkinson's Disease Questionnaire 39 index (0-100 points, higher points indicating worse quality of life) will be determined at baseline and at 6 and 12 months after intervention. The difference between these values will be calculated; Min 0 - Max 100 points (larger decrease indicating stronger improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Scheperjans, MD, Principal Investigator — Helsinki University Central Hospital
Locations (4):
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Päijät-Häme Central Hospital, Lahti
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Yes
Raw sequencing reads will be uploaded to the European Nucleotide Archive. Upon reasonable request and execution of a data transfer agreement we will share de-identified clinical data and metadata in the range that is permitted by local legislation.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After publication of the results for indeterminate time.
Access Criteria: Upon reasonable request and execution of a data transfer agreement.

REFERENCES:
- [Background] Scheperjans F, Levo R, Bosch B, Laaperi M, Pereira PAB, Smolander OP, Aho VTE, Vetkas N, Toivio L, Kainulainen V, Fedorova TD, Lahtinen P, Ortiz R, Kaasinen V, Satokari R, Arkkila P. Fecal Microbiota Transplantation for Treatment of Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2024 Sep 1;81(9):925-938. doi: 10.1001/jamaneurol.2024.2305. PMID 39073834